CLINICAL TRIAL: NCT06375967
Title: Multicenter Study of EUS-guided Gallbladder Drainage vs Choledochoduodenostomy as First Line in Malignant Distal Obstruction in Palliative Patients (CARPEGIEM Trial): an Open-label, Randomized Controlled Clinical Trial
Brief Title: EUS-Gallbladder vs CDS as First Line in MBDO- Palliative (CARPEGIEM Trial)
Acronym: CARPEGIEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other); Hospital General Universitario de Alicante (Other); Hospital Mutua de Terrassa (Other); Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario de Castellón (Other); Complejo Hospitalario de Navarra (Other); University Hospital Virgen de las Nieves (Other); Hospital de Sant Pau (Other); University of Salamanca (Other); Complejo Hospitalario Universitario de Santiago (Other); Complejo Hospitalario Universitario de Vigo (Other)
Responsible Party: Principal Investigator, Joan B Gornals, PhD and Head of Interventional Endoscopy Unit, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARPEGIEM
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-10

CONDITIONS: Malignant Biliary Obstruction; Biliary Tract Neoplasms; Pancreatic Cancer Non-resectable
Keywords: Choledochoduodenostomy; Gallblader drainage; Lumen apposing metal stent; Biliary drainage; Biliopancreatic malignancy
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EUS-GBD with LAMS-Pigtail (Experimental): Biliary drainage using EUS-guided Cholecystostomy with lumen apposing metal stent
  Echoendoscopy-guided Cholecystostomy (EUS-GBD) with deployment of a lumen-apposing metal stent (LAMS) and axis-orienting double-pigtail plastic stent throug LAMS.
  EUS-GBD technique: Diagnostic EUS. Classic or free-hand with preloaded guidewire cholecystostomy with LAMS. Pneumatic dilation whithin LAMS is allowed. 'push' technique'. Deployment of a pigtail coaxial to LAMS.
  Interventions: Procedure: Endoscopic biliary drainage; Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS)
- EUS-CDS with LAMS-Pigtail (Active Comparator): Echoendoscopy-guided Choledochoduodenostomy (EUS-CDS) with deployment of a lumen-apposing metal stent (LAMS) and axis-orienting double-pigtail plastic stent throug LAMS.
  EUS-CDS technique: Diagnostic EUS. Classic or free-hand with preloaded guidewire choledochoduodenostomy with LAMS. Pneumatic dilation whithin LAMS is allowed. In case of bile duct < 15mm is mandatory the 'push' technique. Deployment of a pigtail coaxial to LAMS.
  Interventions: Procedure: Endoscopic biliary drainage; Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS)

INTERVENTIONS:
Procedure: Endoscopic biliary drainage — Decompression of the bile duct by endoscopic aproach.
  Other Names: Biliary drainage
Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS) — Lumen-apposing metal stent (LAMS) with coaxial double-pigtail plastic stent (DPPS) deployment:
  * LAMS size: 6x8mm, 8x8mm. Consider 10x10mm or 10x15mm if abundant pathological material in gallblader.
  * DPPS size: 7Fr x 3-5-7cm.
  Arms: EUS-GBD with LAMS-Pigtail
Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS) — Lumen-apposing metal stent (LAMS) with coaxial double-pigtail plastic stent (DPPS) deployment:
  * LAMS size: 6x8mm or 8x8mm. Consider 10x10mm if bile duct > 18mm.
  * DPPS size: 7Fr x 3-7cm.
  Arms: EUS-CDS with LAMS-Pigtail

SUMMARY:
The aim of the study is to evaluate technical, clinical and safety outcomes of lumen-apposing metal stent (LAMS) with a coaxial double-pigtail plastic stent (DPS) in EUS-guided choledochoduodenostomies vs cholcystogastrostomy for the management of malignant biliary obstruction in palliative patients.

DETAILED DESCRIPTION:
Ecoendoscopy-guided choledochoduodenostomy (EUS-CDS) with a biliary lumen-apposing metal stent (LAMS) has been widely accepted as a second line treatment in cases of ERCP failure in malignant distal biliary obstruction (MDBO). Recent studies (DRAMBO and ELEMENT trial) compared EUS-CDS vs ERCP as a first line treatment in MDBO in palliative patients, showing similar clinical and techinal success and adverse events rate between both techniques, demonstrating that both procedures could be options for primary biliary drainage in unresectable MDBO.

Furthermore a recent clinical trial (BAMPI trial) has proven that the addition of a coaxial double pigtail (DPS) offers benefits in terms of safey and clinical success.

In the last years there has been an increasing interest for the EUS-guided gallblader drainage (EUS-GBD) in unresectable MDBO as an alternative for EUS-CDS, and recent studies and reviews have been reported with acceptable techinal and clinical success, but no clinical trial has been performed up to date.

Our hypothesis is that EUS-GBD may offer benefits in terms of safety over EUS-CDS, maintaining similar clinical and techinal success rates.

ELIGIBILITY:
Inclusion Criteria:

* Malignant distal biliary obstruction diagnosed in patient considered PALIATIVE with biliary drainage indication.
* Consensual malignancy by a bilio-pancreatic multidisciplinar committe (histological confirmation is not mandatory)
* Patient capable of understanding and/or singning the informed consent.
* Patient who understands the type of study and will comply with all follow-up tests throughout its duration

Exclusion Criteria:

* Pregnancy or lactation.
* Severe coagulation disorder: INR > 1.5 non correctable with plasma administration and/or platelet count < 50.000/mm3.
* Previous cholecistectomy or gallblader perforation.
* Tumoral obstruction of cystic duct.
* Multiple liver metastases affecting more than 30% of the liver parenchyma
* Distal malignant biliary strictures in patients considered resectable or borderline.
* Benign or uncertain etiology of biliary strictures or strictures located proximally or in close proximity to the hilum.
* Patients with prior biliary stents or other biliary drainages (e.g., PTCD).
* Altered intestinal anatomy due to prior surgery that prevents or hinders papillary access ______________ (e.g., gastric bypass, Billroth II, duodenal switch, Roux-en-Y).
* Gastric outlet obstruction.
* Situations that do not allow for upper gastrointestinal endoscopy (e.g., esophageal stricture).
* Patients with functional diversity, who lack the capacity to understand the nature and potential consequences of the study, except when a legal representative is available.
* Patients incapable of maintaining follow-up appointments (lack of adherence).
* Lack of informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
RELATED ADVERSE EVENTS | 12 months
  Safety will be measured by careful and comparative evaluation of adverse effects in both groups.
Patients with Recurrent biliary obstruction | 12 months
  Recurrent biliary obstruction (RBO) has been defined as a composite endpoint of either occlusion or migration.

SECONDARY OUTCOMES:
CLINICAL SUCCESS | 2 weeks
  Resolution of jaundice or drop in total bilirubin level by > 50% within 2 weeks after the EUS guided drainage.
TECHNICAL SUCCESS | 24 hours
  Technical success was defined as successful placement of the LAMS between the bile duct (choledoc or gallblader) and the lumen digestive system (stomach or duodenum), creating a transmural ostomy. To evaluate the correct position of the transmural stent, the deployment of the internal flap in the lumen of the bile duct must be verified by ultrasound vision and the internal flap by endoscopic vision.
BILIARY REINTERVENTIONS (BRI) | 12 months
  Interventions needed to treat - Recurrent biliary obstruction (RBO) has been defined as a composite endpoint of either occlusion or migration.
HOSPITAL STAY | 12 months
  Length of hospital stay after intervention
MORTALITY | 12 months
  Overall mortality throughout the study
COST ANALYSIS | 12 months
  Evaluate the costs between the two types of strategy

CONTACTS AND LOCATIONS:
Overall Officials: Joan B Gornals Soler, Principal Investigator — Study Principal Investigator; Carme Loras, Principal Investigator — Hospital Universitari Mutua de Terrassa
Locations (10):
- Spain (10):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, BARCELONA
  - Hospital General Alicante, Alicante, Valencia
  - Hospital Universitari de Castello, Castellon, Valencia
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Virgen de Las Nieves, Granada
  - Complejo Hospitalario de Pamplona, Pamplona
  - Hospital Santiago de Compostela, Santiago de Compostela
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Clinic de Valencia, Valencia
  - Hospital Cunqueiro de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teoh AYB, Napoleon B, Kunda R, Arcidiacono PG, Kongkam P, Larghi A, Van der Merwe S, Jacques J, Legros R, Thawee RE, Saxena P, Aerts M, Archibugi L, Chan SM, Fumex F, Kaffes AJ, Ma MTW, Messaoudi N, Rizzatti G, Ng KKC, Ng EKW, Chiu PWY. EUS-Guided Choledocho-duodenostomy Using Lumen Apposing Stent Versus ERCP With Covered Metallic Stents in Patients With Unresectable Malignant Distal Biliary Obstruction: A Multicenter Randomized Controlled Trial (DRA-MBO Trial). Gastroenterology. 2023 Aug;165(2):473-482.e2. doi: 10.1053/j.gastro.2023.04.016. Epub 2023 Apr 28. PMID 37121331
- [Background] Mangiavillano B, Moon JH, Facciorusso A, Vargas-Madrigal J, Di Matteo F, Rizzatti G, De Luca L, Forti E, Mutignani M, Al-Lehibi A, Paduano D, Bulajic M, Decembrino F, Auriemma F, Franchellucci G, De Marco A, Gentile C, Shin IS, Rea R, Massidda M, Calabrese F, Mirante VG, Ofosu A, Crino SF, Hassan C, Repici A, Larghi A. Endoscopic ultrasound-guided gallbladder drainage as a first approach for jaundice palliation in unresectable malignant distal biliary obstruction: Prospective study. Dig Endosc. 2024 Mar;36(3):351-358. doi: 10.1111/den.14606. Epub 2023 Jul 3. PMID 37253185
- [Background] Binda C, Anderloni A, Fugazza A, Amato A, de Nucci G, Redaelli A, Di Mitri R, Cugia L, Pollino V, Macchiarelli R, Mangiavillano B, Forti E, Brancaccio ML, Badas R, Maida M, Sinagra E, Repici A, Fabbri C, Tarantino I. EUS-guided gallbladder drainage using a lumen-apposing metal stent as rescue treatment for malignant distal biliary obstruction: a large multicenter experience. Gastrointest Endosc. 2023 Nov;98(5):765-773. doi: 10.1016/j.gie.2023.06.054. Epub 2023 Jun 29. PMID 37392954
- [Background] Kamal F, Khan MA, Lee-Smith W, Sharma S, Acharya A, Farooq U, Aziz M, Kouanda A, Dai SC, Munroe CA, Arain M, Adler DG. Efficacy and safety of EUS-guided gallbladder drainage for rescue treatment of malignant biliary obstruction: A systematic review and meta-analysis. Endosc Ultrasound. 2023 Jan-Feb;12(1):8-15. doi: 10.4103/EUS-D-21-00206. PMID 36861505
- [Background] Chen YI, Callichurn K, Chatterjee A, Desilets E, Fergal D, Forbes N, Gan I, Kenshil S, Khashab MA, Kunda R, Lam E, May G, Mohamed R, Mosko J, Paquin SC, Sahai A, Sandha G, Teshima C, Barkun A, Barkun J, Bessissow A, Candido K, Martel M, Miller C, Waschke K, Zogopoulos G, Wong C; ELEMENT trial and for the Canadian Endoscopic Research Collaborative (CERC). ELEMENT TRIAL: study protocol for a randomized controlled trial on endoscopic ultrasound-guided biliary drainage of first intent with a lumen-apposing metal stent vs. endoscopic retrograde cholangio-pancreatography in the management of malignant distal biliary obstruction. Trials. 2019 Dec 9;20(1):696. doi: 10.1186/s13063-019-3918-y. PMID 31818329
- [Background] Garcia-Sumalla A, Loras C, Sanchiz V, Sanz RP, Vazquez-Sequeiros E, Aparicio JR, de la Serna-Higuera C, Luna-Rodriguez D, Andujar X, Capilla M, Barbera T, Foruny-Olcina JR, Martinez B, Dura M, Salord S, Laquente B, Tebe C, Videla S, Perez-Miranda M, Gornals JB; Spanish Working Group on Endoscopic Ultrasound Guided Biliary Drainage. Multicenter study of lumen-apposing metal stents with or without pigtail in endoscopic ultrasound-guided biliary drainage for malignant obstruction-BAMPI TRIAL: an open-label, randomized controlled trial protocol. Trials. 2022 Feb 25;23(1):181. doi: 10.1186/s13063-022-06106-1. Erratum In: Trials. 2022 Mar 14;23(1):214. doi: 10.1186/s13063-022-06138-7. PMID 35216619